CLINICAL TRIAL: NCT03202849
Title: A Randomized Double Blinded Trial of Vitamin D Supplementation With or Without Vitamin A Supplementation in Allogeneic Stem Cell Transplantation
Brief Title: A Randomized Trial of Vitamin D Supplementation With or Without Vitamin A in Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-9480
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: hematopoietic stem cell transplant; vitamin a; vitamin d
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D and A Supplementation (Experimental): Participants receive a single dose of vitamin D and a single dose of vitamin A prior to HSCT.
  Interventions: Dietary Supplement: Vitamin D and A
- Vitamin D Supplementation with Placebo (Active Comparator): Participants receive a single dose of vitamin D and a single dose of placebo prior to HSCT.
  Interventions: Dietary Supplement: Vitamin D and Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D and A — A single dose of Vitamin A and Vitamin D will be given.
  Arms: Vitamin D and A Supplementation
Dietary Supplement: Vitamin D and Placebo — A single dose of Vitamin D plus a placebo will be given.
  Arms: Vitamin D Supplementation with Placebo

SUMMARY:
The investigators hypothesize that supplementation with vitamins A and D will reduce the incidence of acute gastrointestinal graft versus host disease (GI GVHD) compared with supplementation with vitamin D alone.

DETAILED DESCRIPTION:
The investigators' preliminary data suggest that low levels of vitamin A directly impact risk of mucosal barrier injury laboratory-confirmed bloodstream infection (MBI-LCBI) and they believe supplemental vitamin A at the time of hematopoietic stem cell transplantation (HSCT) can reduce the risk of MBI-LCBI and gastrointestinal graft versus host disease (GI GVHD). In addition, the investigators' preliminary data suggest that a significant number of patients requiring HSCT have vitamin D deficiency even prior to transplantation, and that persistent and newly developed deficiency post-HSCT resulted in worse outcomes.

This study is a comparison of vitamin D supplementation comparing a single large dose of vitamin D "stoss therapy" with a placebo in the standard care arm with supplementation with single large doses of both vitamins D and A in the experimental arm. Participants will be randomly assigned to either the standard care arm or the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for allogeneic stem cell transplant
* Vitamin D level < 50 ng/ml
* Vitamin A level < 75th centile for age
* Able to tolerate enteral vitamin dose administration

Exclusion Criteria:

* History of pathologic fractures
* Known history of nephrocalcinosis or nephrolithiasis
* Current granulomatous disease
* ALT > 10X ULN for age prior to administration of vitamin A
* Ongoing raised intracranial pressure
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
GI GVHD | 100 days after transplant
  Incidence of acute GI GVHD at day +100 after transplant. GVHD will be graded by the treating physician as per the modified Glucksberg criteria.

SECONDARY OUTCOMES:
MBI-LCBI | 100 days after transplant
  Incidence of MBI-LCBI at day +100 after transplant.
Treatment Related Mortality | 100 days after transplant
  Treatment related mortality at day +100 after transplant.
Overall Survival | 1 year after transplant
  Overall survival at 1 year after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MBBS, PhD, MRCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khandelwal P, Langenberg L, Luebbering N, Lake KE, Butcher A, Bota K, Ramos KN, Taggart C, Choe H, Vasu S, Teusink-Cross A, Koo J, Wallace G, Romick-Rosendale L, Watanabe-Chailland M, Haslam DB, Lane A, Davies SM. A randomized phase 2 trial of oral vitamin A for graft-versus-host disease in children and young adults. Blood. 2024 Mar 21;143(12):1181-1192. doi: 10.1182/blood.2023022865. PMID 38227933